CLINICAL TRIAL: NCT00565162
Title: A Multicentre, Multinational, Randomised, Open Study to Establish the Optimal Method for Initiating Lantus(Insulin Glargine) Therapy to Determine Metabolic and Economic Outcomes, Safety, and Satisfaction in Subjects With Type 2 Diabetes Mellitus
Brief Title: Insulin Glargine, INITIATE Metabolic and Economic Outcomes of Lantus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4041
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Insulin Glargine — Insulin glargine administered by subcutaneous injection daily at bedtime for 24 weeks.
  Other Names: Lantus

SUMMARY:
To introduce initiation of glargine insulin treatment in primary care based on a patient education program. To show and compare feasibility of group education to individual education program.

ELIGIBILITY:
Inclusion Criteria:

* Insulin-naive Type 2 Diabetes Mellitus subjects, aged ≥18 years and on stable oral anti-diabetic treatment for >6 months requiring basal long-acting insulin (HbA1c >7.5 % and <12.0 %).

Exclusion Criteria:

* The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2003-11; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Superiority is based on observing clinically significant difference in glycaemic control (> than or = to 0,5 % HbA1c). Programs are defined as equally successful if the HbA1c differs less than 0,5 %. | HbA1c values at visits 1, 2, 5 and 10

CONTACTS AND LOCATIONS:
Overall Officials: Sanni Lahdenpera, Study Director — Sanofi
Locations (4):
- Sanofi-Aventis, Helsinki, Finland
- Sanofi-Aventis, Amsterdam, Netherlands
- Sanofi-Aventis, Stockholm, Sweden
- Sanofi-Aventis, Leicester, United Kingdom

REFERENCES:
- [Background] Yki-Jarvinen H, Juurinen L, Alvarsson M, Bystedt T, Caldwell I, Davies M, Lahdenpera S, Nijpels G, Vahatalo M. Initiate Insulin by Aggressive Titration and Education (INITIATE): a randomized study to compare initiation of insulin combination therapy in type 2 diabetic patients individually and in groups. Diabetes Care. 2007 Jun;30(6):1364-9. doi: 10.2337/dc06-1357. Epub 2007 Mar 23. PMID 17384341